CLINICAL TRIAL: NCT05799729
Title: Correlation Between Concentration at the Effector Site of Continuous Infusion of Ketamine (Calculated With DOMINO Pump) and Bispectral Index Values During General Anaesthesia for Breast Surgery
Brief Title: Effect of Ketamine Infusion on BIS Values
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD, Principal investigator, University of Padova
Other Study IDs: KetainfusionMAST
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Anesthesia Brain Monitoring; Ketamine
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CeK 0.1: Data about Continuous infusion with Concentration at the effector site of Ketamine (CeK) set (at anesthesiologist's discretion) at 0.1 ug/ml for at least 30 minute and BIS during a propofol-remifentanil general anesthesia will be correlated.
  Interventions: Drug: Ketamine
- CeK 0.2: Data about Continuous infusion with Concentration at the effector site of Ketamine (CeK) set (at anesthesiologist's discretion) at 0.2 ug/ml for at least 30 minute and BIS during a propofol-remifentanil general anesthesia will be correlated.
  Interventions: Drug: Ketamine
- CeK 0.4: Data about Continuous infusion with Concentration at the effector site of Ketamine (CeK) set (at anesthesiologist's discretion) at 0.4 ug/ml for at least 30 minute and BIS during a propofol-remifentanil general anesthesia will be correlated.
  Interventions: Drug: Ketamine
- CeK 0.6: Data about Continuous infusion with Concentration at the effector site of Ketamine (CeK) set (at anesthesiologist's discretion) at 0.1 ug/ml for at least 30 minute and BIS during a propofol-remifentanil general anesthesia will be correlated.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — CeK will be set at anesthesiologist's discretion. Only patients with continuous infusion of CeK 0.1, 0.2, 0.4 or 0.6 for at least 30 minutes will be considered.

SUMMARY:
Aim of this trial is to define if Concentration at the effector site (Ce) of Ketamine, during a continuous infusion and calculated with DOMINO model infusion pump are correlated with Bispectral Index BIS values during general anaesthesia for breast surgery.

DETAILED DESCRIPTION:
Correlation between Concentration at the effector site (Ce) of Ketamine and Bispectral Index (BIS) values during general anaesthesia for breast surgery has not been defined yet during a continuous infusion.

Authors want to analyze this correlation during general anaesthesia conducted using Propofol, ketamine and remifentanil. All of these drugs will be delivered with Target-Controlled Infusion pumps (in particular Eleveld for Propofol, Minto for Remifentanil and Domino for Ketamine).

Ketamine will be observationally set at anaesthesiologist's discretion, but only CeK 0.1, 0.2, 0.4 and 0.6 for at least 30 minutes will be considered for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Undergo general anaesthesia with Targeted Controlled Infusion of Ketamine (Domino model), Propofol (Schnider model) and Remifentanil (Minto model)

Exclusion Criteria:

* Neurological disease
* Psychiatric disease
* Benzodiazepines intake
* Obesity

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Authors will recruit patients who will undergo breast oncologic surgery and anesthetized with TIVA-TCI propofol,remifentanil and ketamine anesthesia.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Correlation between Concentration at the effector site of Ketamine and BIS values | Data about Drugs concentration and BIS during general anaesthesia will be collected, in particular BIS and TCI Ketamine values during all the duration of anesthesia, from the start of ketamine infusion until the stop of ketamine infusion(30minutes)
  Discover if there is linear correlation between Concentration at the effector site of Ketamine and BIS values during standard general anaesthesia conducted with Propofol, remifenatnil and ketamine delivered with targeted controlled infusion pumps, usually adopted in our Hospital to delivery general anaesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Treviso Regional Hospital, Treviso, TV, Italy

IPD SHARING:
Plan to Share IPD: Undecided